CLINICAL TRIAL: NCT05304767
Title: An Open-label Extension Study to Assess the Long-term Safety and Tolerability of Adjunctive KarXT in Subjects With Inadequately Controlled Symptoms of Schizophrenia
Brief Title: An Extension Study to Assess Long-Term Safety and Tolerability of Adjunctive KarXT in Subjects With Inadequately Controlled Symptoms of Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0009; CN012-0009 (Other: Bristol-Myers Squibb Protocol ID); KAR-013 (Other: Karuna Pharmaceuticals Protocol ID)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug: KarXT (Experimental)
  Interventions: Drug: Xanomeline and Trospium Chloride Capsules

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride Capsules — KarXT 50 mg/20 mg BID KarXT 75mg/20 mg BID KarXT 100mg/20 mg BID KarXT 125mg/30 mg BID

SUMMARY:
This is a Phase 3, multicenter, 52-week, outpatient, open-label extension (OLE) study to evaluate the long-term safety and tolerability of adjunctive KarXT in subjects with schizophrenia with an inadequate response to their current antipsychotic treatment who previously completed the treatment period (Visit 8/Day 42 ± 3) of ARISE Study (KAR-012). The primary objective of the study is to assess the long-term safety and tolerability of adjunctive KarXT (a fixed dose combination of xanomeline and trospium chloride twice daily [BID]) in subjects with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥18 to <66 years at the time of randomization of Study KAR-012
2. Subject has successfully completed the treatment period of Study KAR-012
3. Subject has been compliant with the procedures in Study KAR-012 (in the Investigator's judgement)
4. Subject has been compliant with their background antipsychotic drug in Study KAR-012 in the opinion of the Investigator and based on subject and informant reporting Note: Subjects are required to remain on the same appropriate approved APD as in Study KAR-012 and should stay on that same dose throughout the study.
5. Subject is capable of providing signed Informed Consent Form before any study assessments will be performed
6. Subject resides in a stable living situation, in the opinion of the Investigator
7. Subject has identified a reliable informant/caregiver willing and able to assist with study activities as needed throughout the subject's participation in the study. The informant can complete the study visits assessments via phone (as per local regulations). In Bulgaria, the informant needs to be physically present at all study visits where the Investigator determines that his/her input would be beneficial.
8. Women of childbearing potential (WOCP), or men whose sexual partners are WOCP, must be able and willing to use at least 1 highly effective method of contraception during the study and for at least 1 menstrual cycle (e.g., 30 days) after the last dose of study drug. Sperm donation is not allowed for 30 days after the final dose of the study drug. A female subject is considered to be a WOCP after menarche and until she is in a postmenopausal state for 12 months or otherwise permanently sterile (for which acceptable methods include hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).

Exclusion Criteria:

1. Risk for suicidal behavior during the study as determined by the Investigator's clinical assessment and/or Columbia-Suicide Severity Rating Scale (C-SSRS) as confirmed by the following:

   1. Subject answers "Yes" to "suicidal ideation" Item 4 (active suicidal ideation with some intent to act, without a specific plan) or Item 5 (active suicidal ideation with a specific plan and intent) on the C-SSRS
   2. Non-suicidal self-injurious behavior is not exclusionary
2. Any clinically significant abnormalities, including any finding(s) from ECG, or laboratory test at Visit 6, and the physical examination, vital signs, at the EOT visit of Study KAR-012 that the Investigator, in consultation with the Medical Monitor are considered to jeopardize the safety of the subject
3. Female subject is pregnant
4. If, in the opinion of the Investigator (and/or Sponsor/ Medical Monitor), subject is unsuitable for enrollment in the study or subject has any finding that, in the view of the Investigator (and/or Sponsor /Medical Monitor), may compromise the safety of the subject or affect their ability to adhere to the protocol visit schedule or study requirements
5. Risk of violent or destructive behavior as per Investigator's judgement
6. Subjects participating in another investigational drug or device trial or planning on participating in another clinical trial during the study
7. History or high risk of urinary retention, gastric retention, or narrow angle glaucoma as evaluated by the Investigator
8. Subject is taking, or plans to take while in the study, any prohibited concomitant medication
9. For all male subjects only, any one of the following:

   1. History of bladder stones
   2. History of recurrent urinary tract infections
   3. Serum prostate specific antigen (PSA) >10 ng/mL
   4. An International Prostate Symptom Score (IPSS) of 5 (almost always) on either item 1, 3, 5, or 6
   5. A sum of scores on IPSS items 1, 3, 5, and 6 of ≥9 Note: IPSS will be required only for male subjects ≥ 45 years of age. Subjects already enrolled in the study who do not have available PSA values from Study KAR-012 for baseline value use in Study CN012-0009, will have these assessments at their next clinic visit planned after re-consenting to determine current eligibility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From initial dose to safety follow-up visit (54 weeks) or early termination

SECONDARY OUTCOMES:
Incidence of serious treatment-emergent adverse events (TEAEs) | From initial dose to safety follow-up visit (54 weeks) or early termination
Incidence of TEAEs leading to discontinuation of study drug | From initial dose to safety follow-up visit (54 weeks) or early termination

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (174):
- United States (79):
  - Alea Research, Phoenix, Arizona
  - Pillar Clinical Research LLC, Little Rock, Arkansas
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - CITrials - Bellflower, Bellflower, California
  - Local Institution - 110, Cerritos, California
  - Local Institution - 167, Culver City, California
  - Local Institution - 127, Garden Grove, California
  - Local Institution - 152, La Habra, California
  - Local Institution - 126, Lafayette, California
  - Synergy Clinical Research of Escondido, Lemon Grove, California
  - Local Institution - 141, Los Angeles, California
  - Excell Research, Inc., Oceanside, California
  - NRC Research Institute, Orange, California
  - CNRI - Los Angeles, LLC, Pico Rivera, California
  - CITrials, Inc. - Riverside & San Bernardino County, Riverside, California
  - Local Institution - 193, San Diego, California
  - Local Institution - 164, Stanford, California
  - Local Institution - 109, Torrance, California
  - Prestige Clinical Research Center, Inc., Coral Gables, Florida
  - Reliable Clinical Research LLC, Hialeah, Florida
  - Galiz Research, LLC, Hialeah, Florida
  - Local Institution - 105, Lauderhill, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Local Institution - 171, Miami, Florida
  - Local Institution - 173, Miami Lakes, Florida
  - Local Institution - 120, Miami Lakes, Florida
  - Assertive Research Center, Miami Lakes, Florida
  - Local Institution - 124, Orange City, Florida
  - Pines Care Research Center, Inc., Pembroke Pines, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Local Institution - 111, Atlanta, Georgia
  - CenExel Atlanta Center for Medical Research, Atlanta, Georgia
  - Local Institution - 135, Augusta, Georgia
  - CenExel iResearch Atlanta, Decatur, Georgia
  - Psych Atlanta, P.C., Marietta, Georgia
  - Local Institution - 191, Savannah, Georgia
  - Local Institution - 177, Chicago, Illinois
  - Local Institution - 142, Chicago, Illinois
  - Local Institution - 143, Chicago, Illinois
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Local Institution - 139, Overland Park, Kansas
  - Local Institution - 154, Monroe, Louisiana
  - Local Institution - 166, Gaithersburg, Maryland
  - Local Institution - 158, Boston, Massachusetts
  - Boston University - PARENT, Boston, Massachusetts
  - Local Institution - 269, Boston, Massachusetts
  - Local Institution - 185, Worcester, Massachusetts
  - Local Institution - 184, Ann Arbor, Michigan
  - Local Institution - 149, Grand Rapids, Michigan
  - Local Institution - 162, Kalamazoo, Michigan
  - Local Institution - 129, St Louis, Missouri
  - Arch Clinical Trials LLC, St Louis, Missouri
  - Omaha Insomnia and Psychiatric Services LLC, Omaha, Nebraska
  - Local Institution - 147, Las Vegas, Nevada
  - Local Institution - 148, Las Vegas, Nevada
  - CenExel HRI Marlton, Berlin, New Jersey
  - Local Institution - 104, New York, New York
  - Manhattan Psychiatric Center, New York, New York
  - Local Institution - 157, New York, New York
  - Psychiatry and Alzheimer's Care of Rochester. PLLC, Rochester, New York
  - Richmond Behavioral Associates ERG Clinical Research - New York PLLC, Staten Island, New York
  - Local Institution - 176, Hickory, North Carolina
  - Local Institution - 165, Cincinnati, Ohio
  - Local Institution - 168, Garfield Heights, Ohio
  - Local Institution - 163, Independence, Ohio
  - Local Institution - 194, Oklahoma City, Oklahoma
  - Prevention Science Institute, Eugene, Oregon
  - Community Clinical Research, Inc., Austin, Texas
  - Local Institution - 189, DeSoto, Texas
  - JPS Health Network, Fort Worth, Texas
  - Local Institution - 183, Houston, Texas
  - Clinical Trial Network LLC, Houston, Texas
  - Local Institution - 103, Irving, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - Local Institution - 159, Richmond, Texas
  - Green Mountain Research Institute, Rutland, Vermont
  - Northwest Clinical Research Center, Bellevue, Washington
- Bulgaria (21):
  - Center for Mental Health Center - Sofia District EOOD, Sofia, Sofia-Grad
  - Medical Center Akademika EOOD, Sofia, Sofia-Grad
  - MHAT Dr. Hristo Stambolski, EOOD, Kazanlak, Stara Zagora
  - Ambulatory for Individual Practice for Specialized Medical Care in Psychiatry - Dr Ivo Natsov, Cherven Bryag
  - Local Institution - 311, Dupnitsa
  - Local Institution - 316, Kardzhali
  - State Psychiatric Hospital 'Sv. Ivan Rilski', Novi Iskar, Novi Iskar
  - Medical Center Medconsult Pleven OOD, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT Sv. Georgi, EAD, Plovdiv
  - Local Institution - 321, Plovdiv
  - Local Institution - 313, Razgrad
  - MHAT Dr Ivan Seliminski AD, Sliven
  - Medical Center 'Sv.Naum', Sofia
  - DCC 'Sv. Vrach and Sv. Sv. Kuzma and Damyan', OOD, Sofia
  - Local Institution - 320, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Intermedica, OOD, Sofia
  - Medical Center VAS OOD, Targovishte
  - DCC Mladost M - Varna, OOD, Varna
  - Mental Health Center-Vratsa EOOD, Vratsa
- Czechia (6):
  - Local Institution - 905, Klecany
  - Local Institution - 903, Ostrava - Poruba
  - Local Institution - 904, Pilsen
  - Local Institution - 906, Prague
  - Local Institution - 901, Prague
  - Local Institution - 902, Prague
- India (17):
  - Local Institution - 616, Guwahati, Assam
  - Local Institution - 607, Ahmedabad, Gujarat
  - Local Institution - 604, Ahmedabad, Gujarat
  - Local Institution - 609, Surat, Gujarat
  - Local Institution - 613, Vadodara, Gujarat
  - Local Institution - 617, Belgavi, Karnataka
  - Local Institution - 614, Mangalore, Karnataka
  - Local Institution - 602, Mangalore, Karnataka
  - Local Institution - 601, Mysore, Karnataka
  - Local Institution - 611, Kozhikode, Kerala
  - Local Institution - 610, Aurangabad, Maharashtra
  - Local Institution - 603, Nagpur, Maharashtra
  - Local Institution - 608, Nashik, Maharashtra
  - Local Institution - 605, Nashik, Maharashtra
  - Local Institution - 615, Ajmer, Rajasthan
  - Local Institution - 606, Rajkot, Rajasthan
  - Local Institution - 612, Lucknow, Uttar Pradesh
- Japan (9):
  - Local Institution - 258, Konan-shi, Aichi-ken
  - Local Institution - 250, Toyoake-shi, Aichi-ken
  - Local Institution - 255, Fukuoka, Fukuoka
  - Local Institution - 257, Shirakawa-shi, Fukushima
  - Local Institution - 254, Karatsu-shi, Saga-ken
  - Local Institution - 253, Meguro-ku, Tokyo
  - Sangenjaya Neurology- Psychosomatic Clinic, Setagaya-ku, Tokyo
  - Local Institution - 910, Shibuya-ku, Tokyo
  - Local Institution - 256, Shinjuku-ku, Tokyo-To
- Poland (9):
  - Local Institution - 506, Bialystok
  - Local Institution - 507, Gdansk
  - Local Institution - 509, Grudziądz
  - Local Institution - 502, Katowice
  - Local Institution - 501, Kielce
  - Local Institution - 503, Lodz
  - Local Institution - 505, Lublin
  - Local Institution - 508, Suchy Las
  - Local Institution - 504, Tuszyn
- Romania (10):
  - Local Institution - 803, Brasov
  - Local Institution - 804, Bucharest
  - Local Institution - 810, Bucharest
  - Local Institution - 802, Bucharest
  - Local Institution - 809, Bucharest
  - Local Institution - 807, Bucharest
  - Local Institution - 808, Craiova
  - Local Institution - 801, Galati
  - Local Institution - 806, Iași
  - Local Institution - 805, Sibiu
- Serbia (15):
  - Local Institution - 403, Belgrade
  - Clinical Center ' Dr Dragisa Misovic Dedinje', Belgrade
  - Local Institution - 413, Belgrade
  - Local Institution - 417, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Local Institution - 411, Gornja Toponica
  - Special Hospital for Psychiatric Diseases 'Kovin', Kovin
  - Local Institution - 404, Kovin
  - Local Institution - 406, Kragujevac
  - Local Institution - 408, Kragujevac
  - University Clinical Center Kragujevac, Kragujevac
  - Local Institution - 415, Niš
  - Local Institution - 416, Novi Kneževac
  - Special Hospital for Psychiatric Diseases 'Sveti Vracevi', Novi Kneževac
  - Local Institution - 409, Vršac
- United Kingdom (8):
  - Local Institution - 707, Bodmin, Cornwall
  - Local Institution - 705, Brighton, East Sussex
  - Local Institution - 701, London, Greater London
  - Local Institution - 706, Ashton-under-Lyne, Lancashire
  - Local Institution - 708, Oxford, Oxfordshire
  - Local Institution - 702, Chertsey, Surrey
  - Local Institution - 703, Birmingham, West Midlands
  - Local Institution - 704, Glasgow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05304767.html